CLINICAL TRIAL: NCT00311506
Title: A Study to Determine the Variability of a 6-Minute Walk Test in Cystic Fibrosis Subjects With Advanced Lung Disease
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Other Study IDs: Z1943n
Record Dates: First submitted 2006-03-25; First posted 2006-04-06 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cystic Fibrosis
Keywords: Pulmozyme
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is an observational study to be conducted at approximately 25 sites in the United States. Approximately 25 subjects with severe obstructive CF lung disease (FVC <40% predicted) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Males or females who will be >=14 years old at Visit 3
* A proven diagnosis of CF as evidenced by a positive sweat test (sweat sodium or chloride >60 mEq/L by quantitative pilocarpine iontophoresis), or genotype and clinical symptoms consistent with the diagnosis of CF
* Able to perform reproducible spirometry maneuvers at Visit 1 in accordance with the American Thoracic Society (coefficient of variation for three FEV1 maneuvers <=0.2)
* FVC <40% predicted for height, age and sex at Visit 1
* On a stable regimen of chest physiotherapy (CPT) begun at least 7 days prior to Visit 1
* Able to complete the 6-minute walk test at Visit 1

Exclusion Criteria:

* Use of an investigational drug or device within 28 days prior to Visit 1
* Experiencing an episode of severe acute respiratory failure, as determined by the investigator

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 1999-10 (Actual); Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris Cheeks, M.D., Study Director — Genentech, Inc.